CLINICAL TRIAL: NCT06282588
Title: Treatment of High-Risk Prostate Cancer Guided by Novel Diagnostic Radio- and Molecular Tracers (THUNDER): A Two-part Phase 2/ 3 Trial
Brief Title: Treatment of High-Risk Prostate Cancer Guided by Novel Diagnostic Radio- and Molecular Tracers
Acronym: THUNDER
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cancer Research Antwerp (Other)
Collaborators: Bayer (Industry); Veracyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTO21042GZA
Record Dates: First submitted 2024-01-19; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: High-risk; PSMA PET/CT scan; Decipher
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; Radiotherapy; Goserelin; Drug Implants; Triptorelin Pamoate; Leuprolide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Injections; Docetaxel

STUDY DESIGN:
Intervention Model Description: Phase 2: non randomised, 1 treatment arm, open label Phase 3: randomized 1:1 between two treatment arms, blinded
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Phase 3 trial: blinded Phase 2 trial: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 2 Open Label (Experimental): Darolutamide for up to 96 weeks (24 months) and primary SOC RT
  Interventions: Drug: Darolutamide; Radiation: Radiotherapy
- Phase 3 Blinded Experimental (Experimental): Darolutamide + LHRHA for up to 96 weeks (24 months) and primary SOC RT
  Interventions: Drug: Darolutamide; Radiation: Radiotherapy; Drug: Zoladex 3.6Mg Implant; Drug: Zoladex LA; Drug: Decapeptyl sustained release 22.5 mg; Drug: Decapeptyl sustained release 11.25 mg; Drug: Depo-Eligard 45 mg; Drug: Depo-Eligard 22.5 mg; Drug: Depo-Eligard 7.5 mg; Drug: Firmagon 120 MG Injection; Drug: Firmagon 80 MG Injection; Drug: Docetaxel
- Phase 3 Blinded Comparator (Placebo Comparator): Darolutamide matched placebo + LHRHA for up to 96 weeks (24 months) and primary SOC RT
  Interventions: Drug: Darolutamide matched placebo; Radiation: Radiotherapy; Drug: Zoladex 3.6Mg Implant; Drug: Zoladex LA; Drug: Decapeptyl sustained release 22.5 mg; Drug: Decapeptyl sustained release 11.25 mg; Drug: Depo-Eligard 45 mg; Drug: Depo-Eligard 22.5 mg; Drug: Depo-Eligard 7.5 mg; Drug: Firmagon 120 MG Injection; Drug: Firmagon 80 MG Injection; Drug: Docetaxel

INTERVENTIONS:
Drug: Darolutamide — 2x300 mg tablets twice daily, for up to 96 weeks
  Other Names: Nubeqa; BAY1841788
  Arms: Phase 2 Open Label; Phase 3 Blinded Experimental
Drug: Darolutamide matched placebo — 2x300 mg tablets twice daily, for up to 96 weeks
  Other Names: BAY1841788 matched placebo
  Arms: Phase 3 Blinded Comparator
Radiation: Radiotherapy — Preferred regimens: 60 to 62 Gy delivered in 20 fractions of 3.0 to 3.1Gy per fraction; 36.25 Gy delivered in 5 fractions of 7.25 Gy per fraction, 2-3 fractions per week
Drug: Zoladex 3.6Mg Implant — 3.6 mg, subcutaneous use
  Other Names: Goserelin acetate 3.6 mg
  Arms: Phase 3 Blinded Comparator; Phase 3 Blinded Experimental
Drug: Zoladex LA — 10.8 mg, subcutaneous use
  Other Names: Goserelin acetate 10.8 mg
  Arms: Phase 3 Blinded Comparator; Phase 3 Blinded Experimental
Drug: Decapeptyl sustained release 22.5 mg — 22.5 mg, intramusculair injection
  Other Names: Triptorelin 11.25 mg
  Arms: Phase 3 Blinded Comparator; Phase 3 Blinded Experimental
Drug: Decapeptyl sustained release 11.25 mg — 11.25 mg, intramusculair injection
  Other Names: Triptorelin 11.25 mg
  Arms: Phase 3 Blinded Comparator; Phase 3 Blinded Experimental
Drug: Depo-Eligard 45 mg — 45 mg, subcutaneous use
  Other Names: Leuprorelin acetate 45 mg
  Arms: Phase 3 Blinded Comparator; Phase 3 Blinded Experimental
Drug: Depo-Eligard 22.5 mg — 22.5 mg, subcutaneous use
  Other Names: Leuprorelin acetate 22.5 mg
  Arms: Phase 3 Blinded Comparator; Phase 3 Blinded Experimental
Drug: Depo-Eligard 7.5 mg — 7.5 mg, subcutaneous use
  Other Names: Leuprorelin acetate 7.5 mg
  Arms: Phase 3 Blinded Comparator; Phase 3 Blinded Experimental
Drug: Firmagon 120 MG Injection — 120 mg, subcutaneous use
  Other Names: Degarelix 40 mg
  Arms: Phase 3 Blinded Comparator; Phase 3 Blinded Experimental
Drug: Firmagon 80 MG Injection — 80 mg, subcutaneous use
  Other Names: Degarelix 20 mg
  Arms: Phase 3 Blinded Comparator; Phase 3 Blinded Experimental
Drug: Docetaxel — 75 mg per square m, IV infusion
  Other Names: Taxotere
  Arms: Phase 3 Blinded Comparator; Phase 3 Blinded Experimental

SUMMARY:
This Investigator-initiated, Treatment of High-Risk Prostate Cancer Guided by Novel Diagnostic Radio- and Molecular Tracers (THUNDER) study will be conducted in subjects with high-risk localized or locally advanced prostate cancer (PCa). The study contains both a randomized Phase 3 treatment intensification study, as well as a treatment de-intensification non-randomized Phase 2 study. The aim of the THUNDER study is to improve the outcome of high-risk PCa by improved risk stratification. Novel radiotracers and a genomic classifier (Decipher) will be used to guide treatment decisions, instead of standard imaging which is limited by lower sensitivity and specificity.

The hypothesis for the study is that treatment intensification based on a positive PSMA PET/ CT scan or Decipher high score (> 0.6) improves time to new metastases detected on PSMA PET/ CT in high-risk PCa. In patients who are PSMA PET/ CT negative with a low/ intermediate Decipher score (≤ 0.6), it is hypothesized that treatment de-intensification will improve patient quality of life while maintaining a good oncological outcome.

The study will be conducted at multiple centers across Europe. Participation in the study will comprise a screening period, where the screening assessments must be completed before subjects are enrolled and randomized (only for Phase 3 subjects). Eligible, consenting subjects will then undergo treatment according to their assigned study phase and treatment group, to occur over up to 96 weeks (24 months) with a post-treatment follow-up period to monitor safety and efficacy. The study will be closed when 96 events have been registered for the primary endpoint, which is expected to be at 7-8 years from the time of randomization of the first subject.

DETAILED DESCRIPTION:
Approximately 360 evaluable patients determined to have high-risk localized or locally advanced PCa, with PSMA positive non-localized disease or a Decipher high score (> 0.6) will be enrolled to the Phase 3 trial. Subjects with PSMA positive non-localized disease for which a Decipher result cannot be obtained, will also be enrolled to the Phase 3 study.

All Phase 3 subjects will be randomly assigned in a 1:1 ratio to receive darolutamide plus Luteinizing hormone releasing hormone (ant)-agonists (LHRHA), or darolutamide matched placebo plus LHRHA, for up to 96 weeks (24 months). All Phase 3 subjects will also receive primary standard of care (SOC) radiation therapy (RT). Subjects in Phase 3 should be commenced on an LHRHA and darolutamide or placebo within 14 days after randomization (unless started earlier) plus SOC RT. Only patients with a PSMA PET-CT showing more than 5 M1 lesions are allowed to receive docetaxel in both arms of the Phase 3 trial. Docetaxel should be started within 4 weeks from randomization. Randomization of Phase 3 subjects will be stratified by 1 versus > 1 high-risk features, N1 versus M1 PSMA positive versus PSMA negative disease, Decipher low/ intermediate versus high versus unknown score and clinical trial site.

Approximately 133 evaluable patients determined to have localized PCa by PSMA PET/ CT (PSMA negative) with a low/ intermediate Decipher test score (≤ 0.6) will enter the non-randomized, Phase 2, single treatment arm, de-intensification study. Subjects with localized PCa by PSMA PET/ CT who return a high Decipher score (> 0.6) will be enrolled and randomized into the Phase 3 study. Subjects with localized PCa by PSMA PET/ CT for which a Decipher result cannot be obtained, will be deemed ineligible for study participation.

All Phase 2 study subjects will receive darolutamide for the study duration for up to 96 weeks (24 months) and primary SOC RT.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathology-proven PCa
2. High-risk locally advanced disease is defined as any of the following factors: PSA > 20 ng/mL OR T-stage 3 or 4 OR Gleason score 8-10 OR cN1.

   Note: documentation of the clinical T-stage may be obtained from any clinical assessment acceptable for clinical T staging including physical exam (DRE), transrectal ultrasound, CT or MRI. Documentation for the N1 stage can be defined on CT or MRI.
3. An Eastern Cooperative Oncology Group (ECOG) Performance Status grade of 0 or 1.
4. Willingness to undergo a PSMA PET/ CT with or without contrast.

   1. Subjects who are PSMA PET/ CT positive for at least one regional or distant (extra-pelvic) lesion at screening (PSMA PET scans will be assessed as described in the study imaging manual), will be eligible to be randomized to either arm of the Phase 3 study. A lesion is considered positive if it has a E-PMSA score of 4 or 5.
   2. Pending confirmation of their Decipher score, subjects who are PSMA PET/ CTnegative for regional or distant lesions at screening (PSMA PET scans will be assessed as described in the study imaging manual), will be eligible for inclusion in either the Phase 3 study (if a high [> 0.6] Decipher score is confirmed) or the non-randomized Phase 2 study (if a low/ intermediate [≤ 0.6] Decipher score is confirmed).
5. Willingness to have their primary tumor sequenced for determination of Decipher score

   1. Subjects who have a negative PSMA PET/ CT and a tumor with a low/ intermediate Decipher score (≤ 0.6) will be eligible to enter the non-randomized Phase 2 study.
   2. Subjects who have a negative PSMA PET/ CT and a tumor with a high Decipher score (> 0.6) will be eligible to be randomized to either arm of the Phase 3 study.
   3. In subjects with positive PSMA PET/ CT, the Decipher score will not determine the treatment allocation.
6. Willingness to undergo SOC RT and long-term ADT (treatment with darolutamide and/ or LHRHA)
7. Subject is able and willing to provide written informed consent, which includes compliance with and ability to undergo all study procedures and attend the scheduled follow-up visit/s per protocol.
8. Subject must be over 18 years of age.
9. Subject able to swallow whole study drug tablets.
10. To avoid risk of drug exposure through the ejaculate (even men with vasectomies), subjects must use a condom during sexual activity while on study drug and for 3 months after the last administration of study treatment. Donation of sperm is not allowed during the treatment phase and for 3 months after the last administration of study treatment.
11. Adequate organ function determined by the following local laboratory values:

    1. Adequate bone marrow function: Hemoglobin ≥ 100 g/L, white cell count (WCC) ≥ 4.0 x 109/L, absolute neutrophil count (ANC) ≥ 1.5 x 109/L and platelets > 100 x 109/L
    2. Adequate renal function: calculated creatinine clearance > 30 mL/min (Cockroft-Gault)
    3. Adequate liver function: ALT < 2 x upper limit of normal (ULN) and total bilirubin < 1.5 x ULN, (or if total bilirubin is between 1.5 to 2 x ULN, they must have a normal conjugated bilirubin)
    4. Testosterone levels > 50 ng/dL

Exclusion Criteria:

1. Definitive radiologic evidence of metastatic disease outside of the pelvic nodes (M1a, M1b or M1c) on conventional imaging (i.e., bone scan, CT scan, MRI)
2. PCa with predominant non-adenocarcinoma features (sarcomatoid or spindle or neuroendocrine small cell or squamous cell components or other non-adenocarcinoma)
3. Prior pelvic radiotherapy
4. Contraindications for pelvic radiotherapy
5. Contraindications for ADT (treatment with darolutamide and/ or LHRHA)
6. Contraindications or known allergy to PSMA PET/ CT tracers.
7. Prior local therapy for PCa (e.g., radical prostatectomy, high-intensity focused ultrasound [HIFU], cryotherapy). Subjects with previous transurethral resection of the prostate (TURP) or Millin prostatectomy are eligible for participation
8. Prior systemic therapy for PCa, except for patients with a positive PSMA PET/ CT staging with ADT started no more than 4 weeks prior to randomization.
9. Current use of 5-alpha reductase inhibitor Note: if the alpha reductase inhibitor is stopped ≥ 2 weeks prior to enrollment, the subject is eligible.
10. Current chronic use of opioid analgesics, for ≥3 weeks for oral or ≥7 days for non-oral formulations
11. History of seizure or any condition that may predispose to seizure (including, but not limited to prior stroke, transient ischemic attack or loss of consciousness within ≤1 year prior to enrollment; brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect)
12. Any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the subject
13. Major surgery within 21 days prior to enrollment.
14. History of:

    1. Loss of consciousness or transient ischemic attack or stroke within 6 months prior to enrollment, or
    2. Significant cardiovascular disease within 6 months prior to enrollment: including myocardial infarction, unstable angina, congestive heart failure (New York Heart Association [NYHA] classification Grade 2 or greater), ongoing arrhythmias of Grade > 2 (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] v5.0), thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism), coronary artery bypass graft. Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed.
15. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of darolutamide, including difficulty swallowing tablets
16. History of another malignancy within 5 years prior to enrollment except for those malignancies treated with curative intent with a predicted risk of relapse of less than 10% including but not limited to non-melanoma carcinoma of the skin; or adequately treated, non-muscle-invasive urothelial carcinoma of the bladder (i.e., Tis, Ta and low grade T1 tumors). All such cases with a history of malignancy within the last 5 years are to be discussed with study team before enrollment. Melanoma in-situ and other adequately treated in-situ neoplasms are not considered malignancies for the purposes of eligibility assessment
17. Concurrent illness, including severe infection that might jeopardize the ability of the subject to undergo the procedures outlined in this protocol with reasonable safety (human immunodeficiency virus [HIV] infection is not an exclusion criterion if it is controlled with anti-retroviral drugs that are unaffected by concomitant darolutamide)
18. Subjects who are sexually active with women of childbearing potential and not willing/able to use medically acceptable and highly effective forms of contraception during study treatment and for at least 3 months after the last administration of study treatment. Contraception must include: Additional birth control with low failure rate (less than 1% per year) when used consistently and correctly, e.g., combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device (IUD), intrauterine hormone releasing system (IUS), bilateral tubal occlusion, vasectomized partner, true sexual abstinence.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 3: PSMA PET metastasis free survival (ppMFS) | Time from randomization to the date of at least 1 new PSMA-PET positive distant lesion as compared to baseline or date of death from any cause, assessed up to 42 months
  Improvement in PSMA PET metastasis free survival (ppMFS)
Phase 2: quality of life (sexual subdomain) | At 12 months
  EPIC mean changes in sexual subdomain scores over time will be compared, both for change from baseline and absolute scores
Phase 2: quality of life (hormonal subdomain) | At 12 months
  EPIC mean changes in hormonal subdomain scores over time will be compared, both for change from baseline and absolute scores

SECONDARY OUTCOMES:
Overall survival | Time interval between randomization and time of death, assessed up to 42 months
  Overall survival
Prostate-cancer specific survival | Time interval between randomization and prostate cancer death, assessed up to 42 months
  Prostate-cancer specific survival
Biochemical progression-free survival | Measured from the date of randomization to the date event, or death or censored at the last known follow-up date, assessed up to 42 months
  Increase in PSA of >2 ng/ml above the nadir PSA level
Time to next systemic therapy | Measured from date of randomization to time of death, or censored at the last known follow-up date, assessed up to 42 months
  Time to next systemic therapy
Frequency and severity of adverse events | From signing ICF until 30 days after the last dose of study treatment.
  Frequency and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Piet Ost, MD,PhD, Principal Investigator — Gasthuis Zusters Antwerpen
Locations (11):
- Belgium (11):
  - GZA Sint-Augustinus, Wilrijk, Antwerp
  - OLVZ Aalst, Aalst
  - AZ Sint-Jan, Bruges
  - Saint Luc, Brussels
  - UZA, Edegem
  - UZ Gent, Ghent
  - AZ Sint-Lucas, Ghent
  - AZ Groeninge, Kortrijk
  - CHU Liège, Liège
  - AZ Delta, Roeselare
  - VITAZ, Sint-Niklaas

REFERENCES:
- [Derived] Kleiburg F, Dirix P, Fonteyne V, Bral S, De Troyer B, Sautois B, Lamande M, Liefhooghe N, Grisay G, Meersschout S, Vandermeulen A, Jullian N, Staelens L, Poelaert F, Strijbos M, Verschueren J, Goffin K, Withofs N, Ost P. Stage Migration on Prostate-specific Membrane Antigen Positron Emission Tomography/Computed Tomography in Comparison to Conventional Imaging in Patients with High-risk Prostate Cancer Referred for Radiation Therapy: Results from the Phase 2/3 THUNDER Trial. Eur Urol Oncol. 2025 Oct;8(5):1333-1339. doi: 10.1016/j.euo.2025.08.005. Epub 2025 Sep 25. PMID 40998687